CLINICAL TRIAL: NCT04248894
Title: The Impact of High-intensity Interval Training Versus Moderate Continuous Training on Neurovascular Control in Patients With Heart Failure
Brief Title: Impact of Interval Training on Sympathetic Hyperactivity and Vascular Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SDC: 4070/14/050
Record Dates: First submitted 2020-01-23; First posted 2020-01-30 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity interval training (HIIT) (Experimental): High-intensity interval training (HIIT) = the exercise of high intensity perform on a cycle ergometer, three times per week for 12 weeks, and training sessions were matched for energy expenditure (i.e., an isocaloric energy expenditure of 200 Kcal/session). The intensity of the HIIT session was established based on the HR and workload levels corresponding to 5% above the respiratory compensation point.
  Interventions: Other: Exercise training of High Intensity
- Moderate-intensity continuous training (MICT) (Experimental): Moderate-intensity continuous training (MICT) = the exercise of moderate intensity perform on a cycle ergometer, three times per week for 12 weeks, and training sessions were matched for energy expenditure (i.e., an isocaloric energy expenditure of 200 Kcal/session). The intensity of the MICT session was established based on the HR and workload levels corresponding to anaerobic threshold and respiratory compensation point
  Interventions: Other: Exercise training of Moderate Intensity
- No training (Sham Comparator): The patients are instructed to avoid any regular exercise program or any non-supervised exercise protocol during the study.
  Interventions: Other: Untraining

INTERVENTIONS:
Other: Exercise training of High Intensity — High intensity
  Other Names: Physical exercise
  Arms: High-intensity interval training (HIIT)
Other: Exercise training of Moderate Intensity — Moderate intensity
  Arms: Moderate-intensity continuous training (MICT)
Other: Untraining — Sedentary
  Arms: No training

SUMMARY:
In this study, the investigators are testing the hypothesis that reduction in sympathetic activity would be greater following high-intensity interval training (HIIT) than moderate-intensity continuous training (MICT) and correspond with improvements in peripheral vascular function, and skeletal muscle function in patients with heart failure with reduced ejection fraction (HFrEF).

DETAILED DESCRIPTION:
In this study, the investigators are testing the hypothesis that reductions in sympathetic activity would be greater following high-intensity interval training (HIIT) than moderate-intensity continuous training (MICT) and correspond with improvements in peripheral vascular function, and skeletal muscle function in patients with heart failure with reduced ejection fraction (HFrEF). To test this hypothesis patients with chronic heart failure (30 - 65 years), left ventricular ejection fraction ≤40%, Functional Classes II-III), are being randomized into exercise with HIIT, MICT or no training (NT) three times/week for 12 weeks. Muscle sympathetic nerve activity is assessed by microneurography. Brachial artery flow-mediated dilation (FMD), blood flow and vascular conductance were assessed by ultrasonography. Blood pressure (BP) and heart rate (HR) by are being measured via finger photoplethysmograph and peak oxygen uptake (V̇O2peak) by a cardiopulmonary exercise test on ergometer cycle for leg. Biopsy samples from the lateral vast of the thigh are being collected for analysis of the intracellular mechanisms in the skeletal muscle. Exercise training is being conducted under supervision at the Heart Institute, School of Medicine, University of São Paulo. Both HIIT and MICT are performed on a cycle ergometer, three times per week for 12 weeks, and training sessions were matched for energy expenditure (i.e., an isocaloric energy expenditure of 200 Kcal/session). The intensity of the MICT session is established based on the HR and workload levels corresponding to anaerobic threshold and respiratory compensation point (RCP). The intensity of the HIIT session is established based on the HR and workload levels corresponding to 5% above the RCP. All exercise sessions were performed under the supervision of an exercise physiologist. The patients in the NT group were instructed to avoid any regular exercise program or any non-supervised exercise protocol during the study. All patients are being assessed before (pre) and after (post) both exercise training modes or control, no training.

ELIGIBILITY:
Inclusion Criteria:

* Functional Class II to III of New York Heart Association
* Left ventricular ejection fraction ≤40%
* Peak oxygen uptake (V̇O2) <20 ml•kg-1•min-1

Exclusion Criteria:

* Myocardial infarction within three months
* Unstable angina
* Acute heart failure
* Pacemaker
* Pulmonary disease
* Chronic renal disease
* Peripheral neuropathy
* History of stroke
* Untreated hypo/hyperthyroidism
* Body mass index (BMI) >30 kg/m2
* History of smoking

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in muscle sympathetic nerve activity (MSNA) | Baseline and 12 weeks
  MSNA is being assessed by microneurography
Change muscle mechanoreceptor sensitivity | Baseline and 12 weeks
  The mechanoreceptor sensitivity is being assessed via passive exercise to the leg
Change muscle metaboreceptor sensitivity | Baseline and 12 weeks
  The metaboreceptor sensitivity is being assessed via dynamic exercise to the leg.The exercise intensity is 30% maximum voluntary contraction.
Change in chemoreceptor sensitivity | Baseline and 12 weeks
  Hypoxia via 10% oxygen

SECONDARY OUTCOMES:
Peripheral vascular function | Baseline and 12 weeks
  Brachial artery flow-mediated dilation is being used to assess the vascular function
Skeletal muscle function | Baseline and 12 weeks
  The skeletal muscle function is being assessed in biopsy samples collected in lateral vasts of thigh with needle of biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Calors Negrao, PhD, Principal Investigator — aHeart Institute, University of São Paulo Medical School, São Paulo, Brazil
Locations (2):
- Brazil (2):
  - Heart Institute, São Paulo, Cerqueira Cesar
  - Heart Institute (InCor), São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sales ARK, Azevedo LF, Silva TOC, Rodrigues AG, Oliveira PA, Jordao CP, Andrade ACM, Urias U, Guimaraes GV, Bocchi EA, Alves MJNN, Hajjar LA, Filho RK, Grunewald ZI, Martinez-Lemus LA, Padilla J, Negrao CE. High-Intensity Interval Training Decreases Muscle Sympathetic Nerve Activity and Improves Peripheral Vascular Function in Patients With Heart Failure With Reduced Ejection Fraction. Circ Heart Fail. 2020 Aug;13(8):e007121. doi: 10.1161/CIRCHEARTFAILURE.120.007121. Epub 2020 Jul 16. No abstract available. PMID 32673501
- [Derived] Xiao P, Wang C, Li J, Su H, Yang L, Wu P, Lewno MT, Liu J, Wang X. COP9 Signalosome Suppresses RIPK1-RIPK3-Mediated Cardiomyocyte Necroptosis in Mice. Circ Heart Fail. 2020 Aug;13(8):e006996. doi: 10.1161/CIRCHEARTFAILURE.120.006996. Epub 2020 Jun 24. PMID 32578441